CLINICAL TRIAL: NCT05567848
Title: Accelerated Transcranial Magnetic Stimulation in Psychotic Disorders
Brief Title: Accelerated TMS in Psychosis
Acronym: ATP
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Roscoe Brady, Vice-Chair for Research, Department of Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000689
Record Dates: First submitted 2022-10-01; First posted 2022-10-05 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Prodromal Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizotypal Personality Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- repetitive Transcranial Magnetic Stimulation (rTMS) (Experimental): repetitive Transcranial Magnetic Stimulation (rTMS) in a iTBS pattern to the cerebellum at 100% of resting motor threshold
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS is a technique of TMS that allows the selective external manipulation of neural activity in a non-invasive manner. During TMS, a rapidly changing current is passed through an insulated coil placed against the scalp. This generates a temporary magnetic field that in turn induces electrical current in neurons and allows the modulation of neural circuitry. The combination of TMS with functional MRI allows the selective targeting and modulation of brain networks. The repeated application of rTMS can cause long term changes in behavior and task performance that is reflected in altered brain network connectivity.
  The pattern of rTMS will consist of intermittent Theta Burst Stimulation (iTBS) pattern consisting of 2 s trains of 3 pulses at 50 Hz, repeated at 5 Hz, every 10s for a total of 600 pulses per session. Sessions will be separated by an interval of 50 minutes (up to a total of 8 per day).

SUMMARY:
This study is to determine the tolerability and efficacy of an accelerated schedule of Transcranial Magnetic Stimulation for treating symptoms of psychotic disorders such as schizophrenia.

DETAILED DESCRIPTION:
The aim of this protocol is to test the hypothesis that 'accelerated' Transcranial Magnetic Stimulation (TMS) is safe and efficacious in the treatment of psychotic disorders. TMS is a neuromodulation technique that utilizes magnets to alter neuronal activity non-invasively. TMS has received FDA approval as a therapeutic intervention for multiple psychiatric disorders. Historically, these FDA approved treatments have consisted of daily sessions spread out over multiple weeks. "Accelerated" TMS protocols deliver multiple TMS sessions daily over a shorter time frame (e.g., one week). Evidence from dozens of studies across multiple disorders suggests that these protocols are safe and effective.

In this protocol we will test the hypothesis that a form of TMS previously used to treat symptoms of schizophrenia is safe and effective when delivered on an accelerated schedule. Participants in this trial will receive neuronavigated intermittent theta burst TMS targeted to personalized network targets on an accelerated schedule. Our primary outcomes will be to determine if delivering TMS on this schedule is as safe and easily tolerated as it is in other disorders.

Additional outcomes measured will be to test the impact of accelerated TMS on multiple clinical and cognitive measures as well as neuroimaging markers of symptom response.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Diagnosis of a psychotic disorder (i.e. schizophrenia or schizoaffective disorder) or have been identified as being at clinical high risk for developing a psychotic disorder.
* Must be able to read, speak and understand English
* Must be judged by study staff to be capable of completing the study procedures
* Participants will be in stable outpatient treatment with no recent (within the past 30 days) hospitalizations or changes in their medication regimens.

Exclusion Criteria:

* Diagnostic and Statistical Manual 5 diagnosis of moderate substance use disorder within the past month
* Medications will be reviewed by the PI and a decision about inclusion will be made based on the participant's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination with other central nervous system active drugs. Current published TMS guidelines do not preclude specific medications in the setting of TMS(Rossi et al., 2021)
* Conditions that might result in increased risks of side effects or complications from rTMS or MRI, including:

  * Intracranial pathology from a known genetic disorder (e.g., Neurofibromatosis 1, tuberous sclerosis) or from acquired neurologic disease (e.g. stroke, tumor), cerebral palsy, history of severe head injury, or significant dysmorphology;
  * History of fainting spells of unknown or undetermined etiology that might constitute seizures
  * History of multiple seizures or diagnosis of epilepsy
  * Any progressive (e.g., neurodegenerative) neurological disorder such as multiple sclerosis or Parkinson's disease
  * Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
  * Metal implants (excluding dental fillings) unless cleared by the responsible covering MD (i.e. MRI compatible joint replacement)
  * Pacemaker
  * Implanted medication pump
  * Vagal nerve stimulator
  * Deep brain stimulator or transcutaneous electric nerve stimulation unit
  * Ventriculo-peritoneal shunt
  * Signs of increased intracranial pressure
  * Intracranial lesion
  * History of head injury resulting in prolonged loss of consciousness (>15minutes) or neurological sequelae
  * Pregnancy: All participants capable of becoming pregnant will be required to have a pregnancy test; any participant who is pregnant will not be enrolled in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Tolerability of accelerated TMS | 5 days of multiple session of TMS per day
  Participants will be monitored for routinely surveyed on their experience of side effects of TMS. These include both common effects such as headache or neck pain as well as rarer side effects such as dizziness.

SECONDARY OUTCOMES:
Change in cerebellar-cerebral resting-state functional connectivity | Before treatment (Baseline) and 1 week and 3 weeks post treatment
  Participants will receive a MRI before TMS and after TMS. Resting-state functional MRI data will be collected. Symptom change will be correlated with resting-state functional MRI connectivity change between pre- and post-TMS MRI scans
Change in severity of negative symptoms of schizophrenia | Before treatment (Baseline) and 1 week and 3 weeks and 24 weeks post treatment
  The Positive and Negative Symptoms Scale (PANSS) is a 30-item rating instrument evaluating the presence/absence and severity of positive, negative and general psychopathology of schizophrenia. The scale was developed from the Brief Psychiatric Rating Scale (BPRS) and the Psychopathology Rating Scale. All 30 items are rated on a 7-point scale (1=absent; 7=extreme).
Change in auditory hallucination severity | Before treatment (Baseline) and 1 week and 3 weeks and 24 weeks post treatment
  The Psychotic Symptom Rating Scale, AH subscale (PSYRATS-AH) is an interviewer rated scale to assess auditory hallucination (AH) severity and phenomenology. It measures AH frequency, duration, location, loudness, beliefs regarding origin of voices, amount and degree of negative content of voices, amount and intensity of distress associated with voices, disruption to life caused by voices, and controllability of voices.
Change in information processing speed | Before treatment (Baseline) and 1 week and 3 weeks and 24 weeks post treatment
  The Measurement And Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery (MCCB) is used to provide a relatively brief evaluation of key cognitive domains relevant to schizophrenia and related disorders. It is used as a measure of cognitive change in repeated testing applications.

CONTACTS AND LOCATIONS:
Overall Officials: Roscoe O Brady, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No